CLINICAL TRIAL: NCT01833052
Title: CLaret Embolic Protection ANd TAVI - Trial
Acronym: CLEAN-TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. A. Linke, Prof. Dr. med. A. Linke, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HZL-01-TAVI
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Frequency of Cerebral Perfusion Defects After TAVI; Size of Cerebral Perfusion Defects After TAVI
MeSH Terms: interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Cerebral Protection Filter (Other): Patient is treated with Cerebral protection Filter.
  Interventions: Device: TAVI (Medtronic CoreValve); Device: Claret-Filter
- No Cerebral Protection Filter (Other): Patient is not treated with Cerebral protection Filter.
  Interventions: Device: TAVI (Medtronic CoreValve)

INTERVENTIONS:
Device: TAVI (Medtronic CoreValve)
Device: Claret-Filter
  Arms: Cerebral Protection Filter

SUMMARY:
This prospective, randomized study was designed to investigate the benefit of using a Filter-Protection-Device (Claret MontageTM Dual Filter System) during transcatheter aortic valve implantation (TAVI) with a Medtronic CoreValve®.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be scheduled to undergo an endovascular aortic valve prosthesis (Medtronic CoreValve®) implant procedure with the femoral artery as the intended access site for the valve delivery system.

Exclusion Criteria:

* Patient is unsuitable for TAVI
* Prior Stroke or TIA in the last 12 month
* Carotic stenosis >70%
* Relevant stenosis of the brachiocephalic trunc or the right subclavian artery
* Expected Non-compliance for follow-ups
* Pregnancy
* Patient is already recruited for another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Rate and Size of Cerebral Embolism | 2 days after Intervention
  Primary endpoint ist the rate and the size of cerebral embolism in postinterventional Magnetic Resonance Imaging (MRI).

CONTACTS AND LOCATIONS:
Locations (1):
- Leipzig Herzzentrum, Leipzig, Germany

REFERENCES:
- [Derived] Haussig S, Mangner N, Dwyer MG, Lehmkuhl L, Lucke C, Woitek F, Holzhey DM, Mohr FW, Gutberlet M, Zivadinov R, Schuler G, Linke A. Effect of a Cerebral Protection Device on Brain Lesions Following Transcatheter Aortic Valve Implantation in Patients With Severe Aortic Stenosis: The CLEAN-TAVI Randomized Clinical Trial. JAMA. 2016 Aug 9;316(6):592-601. doi: 10.1001/jama.2016.10302. PMID 27532914